CLINICAL TRIAL: NCT02593825
Title: Efficacy of the START-Play Program for Infants With Neuromotor Disorders
Acronym: START-Play
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duquesne University (Other)
Collaborators: University of Delaware (Other); Virginia Commonwealth University (Other); University of Washington (Other); University of Nebraska Lincoln (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R324A150103
Record Dates: First submitted 2015-10-29; First posted 2015-11-02 (Estimated); Results first posted 2020-09-01 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2023-08

CONDITIONS: Cerebral Palsy; Developmental Delay; Infant Development
MeSH Terms: conditions — Cerebral Palsy; Learning Disabilities | interventions — Commerce; Early Intervention, Educational; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- START-Play intervention (Experimental): Intervention incorporating cognitive factors and focusing on self-initiated movement toward achievement of skill in sitting and reaching to increase problem-solving skills, which will then improve overall developmental outcomes. Visits to home by physical therapist twice weekly with parent training, for 3 months.
  Interventions: Behavioral: START-Play intervention
- Business as Usual (Active Comparator): Early motor intervention provided as standard treatment in the home for infants with motor dysfunction who are just beginning to sit. Dosage and content of intervention may vary from infant to infant and geographically.
  Interventions: Behavioral: Business as usual

INTERVENTIONS:
Behavioral: START-Play intervention — The START-Play group is a perceptual-motor approach, which uses self-initiated goal-directed movements to bolster orienting and attending to objects, while understanding basic relationships of cause and effect through manipulation and focused attention. Generally, activities focus on helping the child attend to significant environmental information, which can be correlated to forces useful for controlling posture and movement. Unlike passive movement therapy, the investigator's approach encourages activity and learning to solve problems linked by movement and manipulation of objects, which then scaffold cognitive skill.
  Other Names: Perceptual motor early intervention for infants
  Arms: START-Play intervention
Behavioral: Business as usual — May include active or passive movement, parent training, positioning, equipment modification, training other team members, functional skill training
  Other Names: Early intervention, physical therapy
  Arms: Business as Usual

SUMMARY:
The purpose of this project is to evaluate the efficacy of Sitting Together And Reaching To Play (START-Play), an intervention designed to target sitting, reaching, and motor-based problem solving to improve development and readiness to learn in infants with motor delays or dysfunction. There is limited research examining the efficacy of early physical intervention on infants with neuromotor dysfunction. In addition, most early motor interventions have not been directly linked to learning, despite the research demonstrating an association between motor activity and cognitive skills. START-Play specifically targets motor skills that lead to greater physical exploration, which has been associated with improved problem solving and global development. A randomized controlled trial of START-Play will be conducted across four states to investigate the impact of the intervention on changes over time in sitting and reaching, subsequent changes in global cognitive development, and the mediating influences of motor skill changes and problem solving. The research team will conduct a randomized controlled trial to evaluate the impact of START-Play on motor development, motor problem solving, global development including cognitive problem solving of infants with neuromotor delay and dysfunction. Infants will experience either the intervention or services as usual for 3 months, with following testing at three time points up until 9 months post intervention. The researchers will determine whether the intervention leads to improved sitting and reaching, which leads to improved motor-based problem solving, which leads to improved global development and problem solving.

DETAILED DESCRIPTION:
Setting: The research will take place in the homes of infants and their families in Pennsylvania, Delaware, Washington, and Virginia.

Sample: There will be approximately 140 infants with neuromotor disorders completing participation in this study, beginning at the age the age of 7 to 16 months, as well as their families and interventionists. Infants will have gross motor delays but be able to sit propped up for at least 3 seconds when they are recruited for participation.

Intervention: Sitting Together And Reaching To Play (START-Play) is an intervention for infants with motor dysfunction or delay in which physical therapists visit the child's home to target work on siting, reaching, and problem solving. The therapist visits the home twice weekly for 3 months. During these visits, therapists and families work together to provide intensive, individualized, daily activities to advance reaching and sitting through small increments of challenge and support for these skills, which then become the building blocks for motor-based problem solving. More specifically, the intervention focuses on self-initiated, goal-directed movements to build orientation and attention to objects, while learning basic relationships of cause and effect. Infants and families in the intervention group will receive this intervention in addition to their usual early intervention services.

Research Design and Methods: This study will use a randomized controlled trial in which infants and their families are randomly assigned to the intervention group (START-Play in addition to usual services) or control group (usual early intervention services), stratified by severity of neuromotor disorder. There will be six measurement sessions during the 12-week intervention period, following by assessments during 1-, 3-, and 9-month follow-up visits. The study aims to determine the efficacy of the intervention on sitting and reaching (proximal outcomes) and motor-based problem solving skills (longer-term proximal outcome), which is hypothesized to serve as mediators to the more distal outcomes of global cognitive development and readiness to learn. The investigators will also explore fidelity of implementation to identify conditions that support fidelity and outcomes, as well as identify other moderating factors related to the child (severity of disorder, health, age, cognitive skill at entry), family (socioeconomic status, home environment), or services (fidelity of implementation, other services provided to child) to explore change over time.

Control Condition: Infants and their families in the control condition will continue to receive their regular Part C early intervention services.

Key Measures: Primary outcome measures in the study include the Gross Motor Function Measure and an observational measure of toy contacts for sitting and reaching, and the Individual and Growth Development Indicators (Early Problem Solving Indicator) and Bayley Scales of Infant and Toddler Development -Third Edition for problem solving and global development. Secondary measures include additional measures of postural control and reaching, child and family characteristics, and fidelity of implementation (logs and checklist).

Data Analytic Strategy: The investigators will use linear mixed modeling (LMM) to determine the efficacy of the intervention on child outcomes. Parallel process growth modeling within a structural equation modeling framework will be used to examine whether improvements in sitting and reaching are mediators leading to improvements in problem solving, which is then a mediator leading to long-term global cognitive development. LMM will also be used to examine moderating variables, as well as secondary motor outcomes.

ELIGIBILITY:
Inclusion Criteria:

* • Infants enter study between 7-16 months of age, when they are able to prop sit for 3 seconds and maintain their head at least to the level of neutral alignment with their trunk.

  * Gross motor delay as reflected in the Bayley III motor subtest >1.0 Standard Deviation below the mean.
  * Neuromotor disorder such as cerebral palsy (CP), or at risk for CP because of extreme prematurity or brain damage that occurred at or around birth, or infants with motor delay of an unspecified origin (no clear diagnosis, but delay as above) -• Minimal movement requirements/Indicators of readiness for change: Sits with support of arms for 3 seconds after being placed. Exhibits at least some spontaneous movement of arms.

Exclusion Criteria:

* • Medical complications that severely limit participation in assessments and intervention such as severe visual and congenital/genetic anomalies, uncontrolled seizure disorder.

  * Diagnosis other than an unchanging neuromotor disorder (examples: autism, Down syndrome, spinal cord injury, acquired head injury, muscle disorder).
  * A child will be excluded if the parents report any of following: 1) if the child has a disability of a progressive nature such as muscular dystrophy; 2) if the child's family plans to move out of the local area within one year from the start of the study; 3) if the child has major surgery planned that might affect physical performance.

Ages: 7 Months to 16 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 134 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2022-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Regina T Harbourne, PhD, Principal Investigator — Duquesne University; Sarah W McCoy, PhD, Principal Investigator — University of Washington; Michele A. Lobo, PhD, Principal Investigator — University of Delaware; Stacey C. Dusing, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Duquesne University, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harbourne RT, Dusing SC, Lobo MA, Westcott-McCoy S, Bovaird J, Sheridan S, Galloway JC, Chang HJ, Hsu LY, Koziol N, Marcinowski EC, Babik I. Sitting Together And Reaching To Play (START-Play): Protocol for a Multisite Randomized Controlled Efficacy Trial on Intervention for Infants With Neuromotor Disorders. Phys Ther. 2018 Jun 1;98(6):494-502. doi: 10.1093/ptj/pzy033. PMID 29767802
- [Derived] Molinini R, Stuyvenburg C, Koziol NA, Harbourne RT, Lobo MA, Willett SL, Bovaird JA, Marcinowski E, Price SK, Shall M, Chu VW, Dusing SC. Developmental Trajectories of Emotional Availability Differ Between Dyads With Children With and Without Motor Delay. Infancy. 2025 May-Jun;30(3):e70027. doi: 10.1111/infa.70027. PMID 40537937
- [Derived] Cunha AB, Babik I, Choi D, Koziol N, Harbourne RT, Dusing SC, McCoy SW, Willett SL, Bovaird JA, Lobo MA. The impact of severity of motor delay, timing of task mastery, and START-play intervention on the development of means-end problem solving in young children. Braz J Phys Ther. 2024 Jan-Feb;28(1):100590. doi: 10.1016/j.bjpt.2024.100590. Epub 2024 Feb 9. PMID 38359542
- [Derived] Koziol NA, Butera CD, Kretch KS, Harbourne RT, Lobo MA, McCoy SW, Hsu LY, Willett SL, Kane AE, Bovaird JA, Dusing SC. Effect of the START-Play Physical Therapy Intervention on Cognitive Skills Depends on Caregiver-Provided Learning Opportunities. Phys Occup Ther Pediatr. 2022;42(5):510-525. doi: 10.1080/01942638.2022.2054301. Epub 2022 Mar 29. PMID 35350970
- [Derived] Harbourne RT, Dusing SC, Lobo MA, McCoy SW, Koziol NA, Hsu LY, Willett S, Marcinowski EC, Babik I, Cunha AB, An M, Chang HJ, Bovaird JA, Sheridan SM. START-Play Physical Therapy Intervention Impacts Motor and Cognitive Outcomes in Infants With Neuromotor Disorders: A Multisite Randomized Clinical Trial. Phys Ther. 2021 Feb 4;101(2):pzaa232. doi: 10.1093/ptj/pzaa232. PMID 33382406
- [Derived] Marcinowski EC, Tripathi T, Hsu LY, Westcott McCoy S, Dusing SC. Sitting skill and the emergence of arms-free sitting affects the frequency of object looking and exploration. Dev Psychobiol. 2019 Nov;61(7):1035-1047. doi: 10.1002/dev.21854. Epub 2019 Apr 22. PMID 31012090

RESULTS

PARTICIPANT FLOW:
Groups:
- START-Play Intervention: Intervention incorporating cognitive factors & focusing on self-initiated movement toward achievement of skill in sitting and reaching to increase problem-solving skills, which will then improve overall developmental outcomes. Visits to home by physical therapist twice weekly with parent training, for 3 months.
  START-Play intervention: The START-Play group is a perceptual-motor approach, which uses self-initiated goal-directed movements to bolster orienting and attending to objects, while understanding basic relationships of cause and effect through manipulation and focused attention. Generally, activities focus on helping the child attend to significant environmental information, which can be correlated to forces useful for controlling posture and movement. Unlike passive movement therapy, the investigator's approach encourages activity and learning to solve problems linked by movement and manipulation of objects, which then scaffold cognitive skill; the focus is not on a "normal
Period: Intervention
Arm/Group | START-Play Intervention | Business as Usual
Started | 67 | 67
Completed | 57 | 55
Not Completed | 10 | 12
Not completed — Lost to Follow-up | 10 | 12
Period: Follow-up
Arm/Group | START-Play Intervention | Business as Usual
Started | 57 | 55
Completed | 57 | 55
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- START-Play: Received the START-Play intervention in addition to their usual early intervention and care
- Business-as-Usual: Received only the usual early intervention and services required due to delays
- Total: Total of all reporting groups
Arm/Group | START-Play | Business-as-Usual | Total
Number analyzed (Participants) | 57 | 55 | 112
Age, Customized [Mean (Standard Deviation); unit: Months]
  Months of age (adjusted for prematurity) | 10.93 (2.63) | 10.67 (2.57) | 10.8 (2.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 26 | 48
  Male | 35 | 29 | 64
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 42 | 37 | 79
  Black | 5 | 6 | 11
  Other | 10 | 12 | 22
Bayley Scales of Infant Development III, Cognitive [Mean (Standard Deviation); unit: units on a scale] — Bayley Infant Scale III; used raw scores to show change over time due to delayed group of infants
  units on a scale | 29.25 (7.14) | 28.4 (6.45) | 28.83 (6.8)

OUTCOME MEASURES:

1. Primary Outcome: Bayley Scales of Infant Development III
Description: Bayley Scales of Infant Development III, cognitive scale; raw scores used to reflect change over time and absolute growth (rather than standard scores) Range: Minimum =20 points; Maximum=60 Higher score = better outcome
Time Frame: Baseline, at end of 3 month intervention, and at 12 months post-baseline
Population: All assessments were video recorded and stored for later scoring by researchers masked to group assignment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | START-Play Intervention | Business as Usual
Number analyzed (Participants) | 57 | 55
score on a scale
  Full group, 3 mo results | 35.9 (7.2) | 33.6 (7.1)
  Severely delayed, 3 mo results: number analyzed (Participants) | 25 | 25
  Severely delayed, 3 mo results | 31.7 (7.7) | 29.4 (6.4)
  Mildly delayed, 3 mo: number analyzed (Participants) | 32 | 30
  Mildly delayed, 3 mo | 39.3 (4.6) | 37.3 (5.4)
  Full group, 12 mo results | 44.63 (12.23) | 43.28 (12.05)
  severly delayed, 12 month: number analyzed (Participants) | 25 | 25
  severly delayed, 12 month | 36.6 (10.94) | 35.11 (10.37)
  mildly delayed, 12 mo: number analyzed (Participants) | 32 | 30
  mildly delayed, 12 mo | 52 (8.06) | 49.95 (8.87)
Statistical Analysis 1: Comparison: START-Play Intervention vs Business as Usual; Also examined these groups in sub-groups of mildly delayed (<2.5 Standard Deviations below the mean on motor Bayley score at baseline) and significantly motor delayed (>2.5 Standard Deviations below the mean on motor Bayley score at baseline); Test type: Superiority — Significance was based on α = .05. Hedges' g, corrected for small sample bias, was calculated as a measure of effect size using the model-predicted group differences in rate of change in the numerator and the pooled standard deviation estimated from the 3 or 12 month assessment (for short- and long-term effects, respectively) in the denominator; p < 0.05, Mixed Models Analysis — Piecewise linear mixed modeling (LMM) was performed to address the study questions. LMM was necessary to account for repeated measures nested within children; Slope = 1.14; Piecewise modeling, using individually-varying timepoints, allowed separate slopes to be estimated across the intervention (baseline to 3 months) and post-intervention (3 to 12 months) phases, and accounted for variation in the time between assessments across children. All models controlled for intercept-level differences by site, as well as intercept- and slope-level differences by baseline-adjusted age and motor severity. Intervention effects were derived via intervention by slope interaction terms. Three-way interaction terms were subsequently added to the models to obtain intervention effects stratified by severity

2. Secondary Outcome: Change in Modified Parent Child Interaction-Dyadic Mini Code
Description: Play and interaction of parent and child, coding of behavior frequency and type of interaction; coded as a total percentage of time the parent provided cognitive opportunities
Time Frame: Baseline, at end of 3 month intervention, and at 6 and 12 months after baseline
Population: caregiver and infants with motor delays
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | START-Play Intervention | Business as Usual
Number analyzed (Participants) | 57 | 55
percentage of time
  Baseline | .22 (.26) | .19 (.22)
  3 months post baseline | .46 (.32) | .34 (.31)
  6 months post baseline | .49 (.32) | .46 (.32)
  12 months post baseline | .65 (.31) | .62 (.30)
Statistical Analysis 1: Comparison: START-Play Intervention vs Business as Usual; Test type: Superiority; p = .05, Linear piecewise modeling; Mean Difference (Final Values) = .192

3. Secondary Outcome: Change in Frequency (Number) of Toy Contacts
Description: behavioral coding of play and hand use, coded from videotape; Coding software used to time contacts during standard reaching task during 5 minute reaching at shoulder level and below.
Time Frame: Baseline, at end of 3 month intervention, and at 12 months after baseline
Population: Compared full group pre and post intervention, and then sub-groups of mild and severe Also examined these groups in sub-groups of mildly delayed (<2.5 Standard Deviations below the mean on motor Bayley score at baseline) and significantly motor delayed (>2.5SD below the mean on motor Bayley score at baseline)
Measure: Mean (Standard Deviation); unit: occurrences
Arm/Group | START-Play | Business-as-Usual
Number analyzed (Participants) | 57 | 55
occurrences
  Full group, 3 mo results | 13.1 (8.7) | 13 (7.9)
  Severely delayed, 3 mo results: number analyzed (Participants) | 24 | 26
  Severely delayed, 3 mo results | 7.2 (4.8) | 9.3 (7.5)
  Mildly delayed, 3 mo: number analyzed (Participants) | 33 | 29
  Mildly delayed, 3 mo | 18.2 (8) | 16.5 (6.7)
  Full group, 12 months | 16.46 (9.48) | 15.03 (8.93)
  severly delayed, 12 month: number analyzed (Participants) | 25 | 25
  severly delayed, 12 month | 13.64 (10.98) | 9.78 (7.26)
  mildly delayed, 12 months: number analyzed (Participants) | 32 | 30
  mildly delayed, 12 months | 19.43 (6.65) | 20.28 (7.3)
Statistical Analysis 1: Comparison: START-Play vs Business-as-Usual; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.05, Mixed Models Analysis; Slope = .92, Standard Error of Mean 0.47 — data shown is for the 12 month time point for the severely delayed group comparison

4. Secondary Outcome: Change in Duration (Time) of Toy Contacts
Description: coding number seconds of videotaped hand use during play; timing coded in a video coding software for behavioral analysis Higher score=better
Time Frame: Baseline, at end of 3 month intervention, and at 12 months after baseline
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | START-Play Intervention | Business as Usual
Number analyzed (Participants) | 57 | 55
seconds
  Baseline | 38.20 (30.88) | 42.28 (30.70)
  3 months post baseline | 44.93 (29.84) | 47.38 (28.88)
  12 months post baseline | 46.87 (28.25) | 44.35 (26.36)

5. Secondary Outcome: Change in Gross Motor Function Measure, Sitting Subscale
Description: Gross motor skills in the sitting subsection of the Gross Motor Function Measure (GMFM) Minimum value=4 Maximum value=60 Higher scores=better outcome
Time Frame: Baseline, at end of 3 month intervention, and at 12 months after baseline
Population: Analyzed full group, and separately the mildly delayed group and the significantly delayed group
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | START-Play | Business-as-Usual
Number analyzed (Participants) | 57 | 55
score on a scale
  Full group, 3 mo results | 35 (14.2) | 31.3 (14.7)
  Severely delayed, 3 mo results: number analyzed (Participants) | 30 | 25
  Severely delayed, 3 mo results | 26.3 (13) | 20.9 (9.5)
  Mildly delayed, 3 mo: number analyzed (Participants) | 27 | 30
  Mildly delayed, 3 mo | 41.9 (10.9) | 40.6 (12.1)
  Full group, 12 mo results | 47.13 (15.95) | 44.88 (17.54)
  severely delayed, 12 month: number analyzed (Participants) | 25 | 25
  severely delayed, 12 month | 38.26 (18.37) | 32.72 (19.72)
  mildly delayed, 12 mo: number analyzed (Participants) | 32 | 30
  mildly delayed, 12 mo | 55.28 (6.63) | 54.39 (6.58)
Statistical Analysis 1: Comparison: START-Play vs Business-as-Usual; Also examined these groups in sub-groups of mildly delayed (<2.5SD below the mean on motor Bayley score at baseline) and significantly motor delayed (>2.5SD below the mean on motor Bayley score at baseline); Test type: Superiority; p < 0.05, Mixed Models Analysis; Slope = 1.02; LMM was necessary to account for repeated measures nested within children. Piecewise modeling, using individually-varying timepoints, allowed separate slopes to be estimated across the intervention (baseline to 3 months)

6. Secondary Outcome: Change in Early Problem Solving Indicator (EPSI)
Description: Infant growth and development indicator of problem solving skills, adapted for children with motor deficits Modified to Assessment of Problem-Solving in Play (APSP) Minimum=30 Maximum=120 Higher=better outcome
Time Frame: Baseline, at end of 3 month intervention, and at 6 and 12 months after baseline
Population: Compared full group and also sub-groups of mild or severely delayed children separately
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | START-Play | Business-as-Usual
Number analyzed (Participants) | 57 | 55
score on a scale
  Full group, 3 mo results | 64.5 (27.9) | 59.2 (30.4)
  Severely delayed, 3 mo results: number analyzed (Participants) | 25 | 25
  Severely delayed, 3 mo results | 57.7 (31.1) | 46.9 (30.9)
  Mildly delayed, 3 mo: number analyzed (Participants) | 32 | 30
  Mildly delayed, 3 mo | 70 (24.3) | 70.2 (25.9)
  Full group, 12 mo results | 90.71 (42.66) | 81.95 (41.92)
  severely delayed, 12 month: number analyzed (Participants) | 25 | 25
  severely delayed, 12 month | 71.98 (41.6) | 61.92 (42.67)
  mildly delayed, 12 mo: number analyzed (Participants) | 32 | 30
  mildly delayed, 12 mo | 107.95 (36.5) | 97.63 (34.68)
Statistical Analysis 1: Comparison: START-Play vs Business-as-Usual; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p < 0.05, Mixed Models Analysis; Slope = 8.70; Piecewise modeling, using individually-varying timepoints, allowed separate slopes to be estimated across the intervention (baseline to 3 months)

7. Secondary Outcome: Change in Reaching (Change in Looking and Hand Contact of Toy)
Description: Looking while contacting toy, frequency of either unimanual or bimanual contact while looking at toy
Time Frame: Baseline, at end of 3 month intervention, and at 12 months after baseline
Population: infants with severe motor delays
Measure: Mean (Standard Deviation); unit: occurrences
Arm/Group | START-Play Intervention | Business as Usual
Number analyzed (Participants) | 25 | 25
occurrences
  Baseline | 4.06 (.88) | 5.96 (1.81)
  3 months post baseline | 7.45 (1.21) | 7.14 (1.48)
  12 months post baseline | 10.83 (1.99) | 7.69 (2.56)
Statistical Analysis 1: Comparison: START-Play Intervention vs Business as Usual; Test type: Superiority; p = 0.417, Mixed Models Analysis; Mean Difference (Final Values) = .01

8. Other Pre Specified Outcome: Change in Postural Measure of Trunk Angle
Description: Angle of forward trunk lean in sitting position
Time Frame: Change over 3 months
Population: Infants with severe delays
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | START-Play Intervention | Business as Usual
Number analyzed (Participants) | 25 | 25
degrees | 10.93 (10.93) | 11.64 (8.23)

ADVERSE EVENTS:
Time Frame: 1 year - while infants were in both intervention phase and at follow-up
Description: Any reporting of injury by therapist or parent
Arm/Group | START-Play | Business-as-Usual
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/55
Other Adverse Events (participants affected / at risk) | 0/57 | 0/55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-07-17): https://cdn.clinicaltrials.gov/large-docs/25/NCT02593825/Prot_000.pdf
  • Statistical Analysis Plan (2015-07-17): https://cdn.clinicaltrials.gov/large-docs/25/NCT02593825/SAP_001.pdf